CLINICAL TRIAL: NCT00000537
Title: Stress Reduction & CVD Morbidity and Mortality in Blacks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 80
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Meditation

INTERVENTIONS:
Behavioral: meditation
Behavioral: relaxation

SUMMARY:
To compare the effects of two stress reduction techniques, Transcendental Meditation (TM) and Progressive Muscle Relaxation (PMR), on the control of mild hypertension in elderly Blacks with hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

Life expectancy for Black Americans is about 10 percent less than for whites. The leading cause of excessive mortality in older Blacks is cardiovascular disease which may be largely due to disproportionately high rates of hypertension in older Blacks. Conventional antihypertensive drug therapies are frequently associated with adverse effects on quality-of-life (QL) and low compliance rates, especially in elderly minority populations.

The present study is an extension of a pilot study on a comparable sample of 80 Black elderly. The previous study, which was the first of its kind, yielded results which indicated that both TM and PMR produced moderate reductions in systolic and diastolic blood pressure, with TM producing the most significant improvements in blood pressure and in quality-of-life. Dr. Schneider hypothesized from this and related evidence that TM should prove to be an effective therapeutic adjunct to regular pharmacotherapy for mild hypertension in elderly Blacks, and should prove even more effective in fostering compliance and in improving overall quality-of-life without any of the unpleasant side effects of anti-hypertensive medications.

DESIGN NARRATIVE:

Randomized. Over an 18-month period, 213 people were screened for inclusion in the study. Of these, 127 with initial diastolic blood pressure of 90 to 109 mm Hg, systolic blood pressure of 189 mm Hg or less, and final baseline blood pressure of 179/104 or less mm Hg were randomized to treatment. Of the 127 participants, 16 did not complete follow-up blood pressure measurements. Thus, 111 subjects completed the study. All subjects were pretested over a four session baseline period on clinic blood pressure, ambulatory blood pressure, cardiovascular and emotional reactivity, and quality-of-life measures. Subjects were then randomly assigned, 36 to TM, 37 to PMR, and 38 to lifestyle modification education control and followed monthly with major post-tests at three months and eighteen months on these variables. The primary outcome variables were changes in clinic systolic and diastolic blood pressure values measured blindly. The secondary outcomes were changes in self-monitored home blood pressure and compliance.

The study was extended through July, 2007 for an additional 5 years of followup of the cohort.

ELIGIBILITY:
Inner-city Blacks with mild hypertension

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schneider — Maharishi International University

REFERENCES:
- [Background] Schneider RH, Staggers F, Alxander CN, Sheppard W, Rainforth M, Kondwani K, Smith S, King CG. A randomised controlled trial of stress reduction for hypertension in older African Americans. Hypertension. 1995 Nov;26(5):820-7. doi: 10.1161/01.hyp.26.5.820. PMID 7591024
- [Background] Alexander CN, Schneider RH, Staggers F, Sheppard W, Clayborne BM, Rainforth M, Salerno J, Kondwani K, Smith S, Walton KG, Egan B. Trial of stress reduction for hypertension in older African Americans. II. Sex and risk subgroup analysis. Hypertension. 1996 Aug;28(2):228-37. doi: 10.1161/01.hyp.28.2.228. PMID 8707387
- [Background] Barnes V, Schneider R, Alexander C, Staggers F. Stress, stress reduction, and hypertension in African Americans: an updated review. J Natl Med Assoc. 1997 Jul;89(7):464-76. PMID 9220696
- [Background] Schneider RH, Alexander CN, Staggers F, Orme-Johnson DW, Rainforth M, Salerno JW, Sheppard W, Castillo-Richmond A, Barnes VA, Nidich SI. A randomized controlled trial of stress reduction in African Americans treated for hypertension for over one year. Am J Hypertens. 2005 Jan;18(1):88-98. doi: 10.1016/j.amjhyper.2004.08.027. PMID 15691622